CLINICAL TRIAL: NCT02451787
Title: The 'Hidden' Biological Impact of Vitamin D Deficiency: a Biomarker Study
Brief Title: The 'Hidden' Biological Impact of Vitamin D Deficiency: a Biomarker Study; Part 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Iris BENZIE, Chair Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Vit D Study part 2 v.1
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): vitamin D supplementation group (2500 IU day for 3 months)
  Interventions: Dietary Supplement: Vitamin D
- Control (Placebo Comparator): no vitamin D supplementation
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 2400 units per day for 3 months
  Other Names: cholecalciferol

SUMMARY:
The investigators major aims are to: determine the vitamin D status of a group of young, apparently healthy adults in Hong Kong; examine inter-relationships between vitamin D status and biomarkers of DNA damage and repair, oxidative stress, inflammation and endothelial health; and, in part 2 of the study, investigate effects of improvement in vitamin D status on these biomarkers and other measures of well-being in those young adults shown to be deficient in vitamin D.

DETAILED DESCRIPTION:
In this part 2 of the study the investigators will investigate the effect of vitamin D supplementation on biomarkers of these 'hidden' changes in apparently healthy young adults. The investigators will also explore the effect of improvement in vitamin D status in young apparently healthy adults in regard to muscular strength and response time, glucose control, a hormone that is linked to vitamin D (parathyroid hormone (PTH) ) and mood.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy, non-smokers
* non-obese
* found (in part1) to have low vitamin D status

Exclusion Criteria:

* chronic illness
* serious illness requiring medical treatment in previous 6 months
* pregnancy
* on regular medication or taking supplements on a regular basis

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
biomarkers of oxidative stress | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Iris F Benzie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No